CLINICAL TRIAL: NCT01344642
Title: Qualitative and Quantitative HIV RNA Detection in Saliva Using the Oragene RNA Kit
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: DNA Genotek (has supplied the kits) (Unknown)
Responsible Party: Curtis Cooper, OHRI
Other Study IDs: 2007614-01H
Record Dates: First submitted 2008-04-21; First posted 2011-04-29 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2008-10

CONDITIONS: HIV Infections
Keywords: HIV; RNA
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if the Oragene.RNA kit is able to detect HIV RNA in saliva.

DETAILED DESCRIPTION:
There is an important need for a rapid, non-invasive, sensitive and specific method for detection of HIV RNA, particularly in clinical settings in which patients at risk for HIV exposure are assessed and screened. A rapid and non-invasive method for quantitative testing of HIV RNA would be also valuable to monitor suppression of HIV RNA as a primary surrogate marker of combination antiretroviral therapy efficacy. An Ottawa-based biotech company (DNA Genotek Inc) has developed and sells to research and clinical labs world-wide a kit (Oragene� DNA Self-collection kit) that permits the collection, stabilization at room temperature, and purification of DNA present in saliva. They have recently developed a kit (Oragene��RNA) that is purported to stabilize RNA in saliva, a non-invasive source of a biological fluid.

ELIGIBILITY:
Inclusion Criteria:

* Four groups of 10 patients each will be recruited:

  * Controls (HIV and HCV seronegative by previous testing)
  * HIV seropositive with HIV RNA >1000 copies/mL and not on combination antiretroviral therapy. No concurrent HCV infection.
  * HIV seropositive with HIV RNA <50 copies/mL as a consequence of combination antiretroviral therapy use. No concurrent HCV infection.
  * HIV seropositive with HIV RNA >1000 copies/mL and not on combination antiretroviral therapy. HCV RNA positive and not on antiviral therapy.

Exclusion Criteria:

* Not fitting one of the 4 groups

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV monoinfected HIV-HCV co-infected HIV and HCV uninfected control
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-10; Primary Completion 2008-05 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa Hospital, General Campus, Ottawa, Ontario, Canada